CLINICAL TRIAL: NCT02138565
Title: Effect of Bariatric Surgery on Kidney Function
Acronym: GAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Peter Rossing, Professor, Steno Diabetes Center Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3005
Record Dates: First submitted 2014-03-24; First posted 2014-05-14 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Obese Subjects Who Will Undergo Gastric By-pass Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bariatric surgery (Experimental)
  Interventions: Procedure: Gastric by-pass surgery

INTERVENTIONS:
Procedure: Gastric by-pass surgery

SUMMARY:
Primary hypothesis:

A large reduction in weight is not associated with a change in accurately measured glomerular filtration rate (GFR) (51Chromium ethylenediaminetetraacetic acid plasma clearance (51Cr-EDTA)).

Secondary hypothesis:

A large reduction in weight is associated with a greater change in estimated GFR (The Modification of Diet in Renal Disease (MDRD-formula)) than in accurately measured GFR.

Other formulas for estimated GFR (Cockcroft Gault, Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI), CKD-EPI with cystatin C) are better correlated with accurately measured GFR.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, older than 18 years of age
* Appointed to gastric by-pass surgery on Hvidovre Hospital, Denmark

Exclusion Criteria:

* Withdrawal of surgical indication
* Severe oedema or ascites

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in accurately measured GFR | Up to 6 months and 18 months after surgery

SECONDARY OUTCOMES:
Change in estimated GFR (as measured by the MDRD formula, the Cockcroft Gault formula, CKD-EPI formula and CKD-EPI with cystatin C formula). | Up to 6 months and 18 months after surgery
Change in 24hour blood pressure | Up to 6 months and 18 months after surgery
Change in arterial stiffness (as measured by sphygmocor) | Up to 6 months and 18 months after surgery
Change in body composition, as measured by Dual-energy X-ray absorptiometry scan (DXA-scan) | Up to 6 months and 18 months after surgery
Change in accurately measured GFR compared with change in estimated GFR | Up to 6 months and 18 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, Professor, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Peter Rossing, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] von Scholten BJ, Persson F, Svane MS, Hansen TW, Madsbad S, Rossing P. Effect of large weight reductions on measured and estimated kidney function. BMC Nephrol. 2017 Feb 6;18(1):52. doi: 10.1186/s12882-017-0474-0. PMID 28166744